CLINICAL TRIAL: NCT04949932
Title: Application of Poly-herbal Powder for Treating Acne Vulgaris: A Randomized, Double-Blind, Placebo-controlled Trial
Brief Title: Application of Poly-herbal Powder for Treating Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Md. Shahab Uddin (Other)
Responsible Party: Sponsor-Investigator, Dr. Md. Shahab Uddin, Principal Investigator, Hamdard University
Organization: Hamdard University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUBREC/2021/09/02
Record Dates: First submitted 2021-06-20; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
Keywords: Poly-herbal; Acne vulgaris; Powder; RCT; Bangladesh
MeSH Terms: conditions — Acne Vulgaris | interventions — turmeric extract; fenugreek seed meal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Poly herbal powder (PHP)
  Interventions: Other: Mixed powder of Lens culinaris, Curcuma longa, Mentha arvensis, Azadirachta indica, and Trigonella foenumgraecum.
- Placebo Arm (Placebo Comparator): Powder of Cicer arietinum
  Interventions: Other: Cicer arietinum powder

INTERVENTIONS:
Other: Mixed powder of Lens culinaris, Curcuma longa, Mentha arvensis, Azadirachta indica, and Trigonella foenumgraecum. — Study subjects were prescribed either PHP or placebo once daily at night for 3 weeks consecutively. A dose of 1-2 tea spoonfuls powder had to mixed with water to make paste. Then it was applied on face (except around the eyes) and had to wait for 20-30 minutes until it dries.Then they were washed face by using normal water.
  Arms: Intervention Arm
Other: Cicer arietinum powder — Study subjects were prescribed either PHP or placebo once daily at night for 3 weeks consecutively. A dose of 1-2 tea spoonfuls powder had to mixed with water to make paste. Then it was applied on face (except around the eyes) and had to wait for 20-30 minutes until it dries.Then they were washed face by using normal water.
  Arms: Placebo Arm

SUMMARY:
Acne is a common problem in adolescence to young adult. But there is no such remedy available for acne treatment which has no side effects. Different types of herbs powder has been using in patients with acne vulgaris in the traditional practice of Indian subcontinent as single form or compound. Scientific evidence have shown many herbs has no known side effects and effective on acne. These herbs have antibacterial, anti-inflammatory and anti-oxidant effects.

So, This study is intended to find out an inexpensive and safe alternative by using some common herbs such as Azadirachta indica, Curcuma longa, Lens culinaris Mentha arvensis and Trigonella foenum-graecum. The aim of the study is to evaluate the clinical efficacy of Poly herbal powder (PHP) for treating patients with acne vulgaris.

Total of 42 adults with acne vulgaris was recruited for this study. Study subjects was included both of male and female with age limit of 18 to 35 years.

Duration of study is 05 months with "day one advertisement" for screening followed by randomization for the treatment. The duration of active participation of each study subject was 3 consecutive weeks or 21days.

Difference of baseline and post intervention mean by Total lesion Count (TLC) compared with placebo and assesses the % of reduction of acne based on The Global Acne Grading System (GAGS) score.

Safety assessment was obtained from the incidence and type of adverse events during study period.

DETAILED DESCRIPTION:
Background:

Due to increasing interest from acne patients concerned about the side effects associated with conventional therapies, complementary and alternative medicine (CAM) has been suggested as a new therapeutic modality for acne vulgaris. Herbal medicine is one of these CAM treatments. Different types of herbs powder has been using in patients with acne vulgaris in the traditional practice of Indian subcontinent as single form or compound. As for example, Azadirachta indica, Curcuma longa, Ocimum sanctum, Lens culinaris, Trigonella foenum-graecum and Mentha arvensis etc. These herbs have antibacterial, anti-inflammatory and anti-oxidant effects. Therefore, this study was designed to evaluate the efficacy of poly-herbal powder (PHP) for treating acne vulgaris using some of these plants.

Objective:

To evaluate the clinical efficacy of PHP compared with that of placebo (PBO) in patients with acne vulgaris.

Sample Size:

Literature review have shown that sample size were included 20, 40, 75 and 503 study subjects in various research for treating acne vulgaris. Prior study has shown that the mean±SD of acne vulgaris at the baseline was 19.66 ±3.93 and after intervention it was 14.33±5.96 according to GAGS. Based on this results, the estimated enrollment of 15 per treatment group among those with acne vulgaris would provide the study with a statistical power of 80% (α = 0.05) and Confidence interval of 95% to detect the significant efficacy in acne. By using OpenEpi online calculator, required sample size is 30. But possibility of loss to follow up the inflated sample size is 42.

Methods:

For study subjects recruitment, advertisement was posted on online social networking platforms (such as facebook, Facebook Messenger, facebook groups, linkedIn, what's up and e-mail). The all relevant study requirements was included in the advertisement following a link of Google Form Questionnaire (socio-demographic data, specially instructed photograph) to participate in this study. Enrollment of respondent was done by acne lesions counting from the photograph sent by the study subjects through Google Form following fulfillment of inclusion criteria.

Thereafter, Study subject was assigned to either PHP or PBO randomly for 03 consecutive weeks and intervention products was sent by courier according to study subject's present address. After intervention period study subjects was had to fill another Google Form Questionnaire including socio-demographic data, specially instructed photograph and other information.

(Instructions for Taking Photograph: Mobile phone with camera, camera resolution must be 8 or more than 8 Mega pixels. Study subject has to take photo from a distance of 12 inches from face. Upload total of 6 photos (Right sided 2 photos, Left sided 2 photos and 2 photos from front) of face.)

An intention-to-treat analysis will be conducted for patients who have received intervention at least once. Data will be presented as mean±SD and percentage of reduction in the change of counting acne lesions with 95% confidence interval and p=0.05.

Efficacy Assessment:

Difference of baseline and post intervention mean by Total lesion Count (TLC) compared with placebo and assesses the % of reduction of acne based on GAGS score. Difference between two means will be compared with independent two sample t-test.

The Global Acne Grading System (GAGS):

The GAGS is a quantitative scoring system to assess acne severity. It was first developed by Doshi and colleagues in 1997. The total severity score is derived from summation of six regional sub scores. Each is derived by multiplying the factors-2 for forehead, 2 for each check, 1 for nose, 1 for chin, 3 for both chest and back by the most heavily weighted lesion within each region (1 for ≥ one comedone, 2 for ≥ one papule,3 for ≥ one pustule, and 4 for ≥ one nodule). The regional factors were derived from consideration of surface area and distribution and density of pilosebaceous units. The summation of local score indicates, "0 = None, 1-18 = Mild, 19-30 = Moderate, 31-38 = Severe, > 39 = Very severe."

Data and Safety Monitoring:

To maintain the quality of this trial, data & safety monitoring will be conducted by Data & Safety Monitoring Board (DSMB). The members of the DSMB was included that individual who was not involved directly in this research. For this clinical trial, DSMB members was joined from the Faculty of Unani and Ayurvedic Medicine of Hamdard University Bangladesh (HUB).

Safety assessment was obtained from the incidence and type of adverse events during study period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women both aged between 18-35 years
* Presenting minimum 5 acne lesions (whiteheads, blackheads, papules, pustules, nodules)
* Study subject who will be agreed with Online informed consent.

Exclusion Criteria:

* Have infected acne lesions
* If study subject suffers from any serious medical conditions such as uncontrolled hypertension, diabetes mellitus, past or current malignancy, liver or kidney dysfunction, active pulmonary tuberculosis other severe dermatitis, or any infectious or systemic diseases.
* Use of a topical medication containing steroids for the treatment of skin disease more than once per month.
* Hypersensitive skin.
* Erythema, or telangiectasia at the test site.
* Use of the same or similar cosmetics (or pharmaceutical) on the test site within three months of screening.
* Having undergone a skin peeling or having wrinkles removed within six months.
* Any other reasons of unsuitability for the clinical trial at the discretion of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Lesions Count (TLC) | 03 weeks
  Total Lesions Count (TLC) = Comedones + Papules + Pastules, before and after intervention will be presented as percentage as well as mean and standard deviation.

SECONDARY OUTCOMES:
Change in The Global Acne Grading System score | 03 weeks
  The total severity score is derived from summation of six regional (i.e forehead, check, nose, chin, chest and back) sub scores. The summation of local score indicates, "0 = None, 1-18 = Mild, 19-30 = Moderate, 31-38 = Severe, > 39 = Very severe."
Change in non-inflammatory and inflammatory lesions count | 03 weeks
  Pre and post treatment changes in non-inflammatory ( i.e Comedones) and inflammatory (i.e papule, pustule & nodule) acne lesions count will be presented as percentage as well as mean and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Md. S Uddin, BUMS, Principal Investigator — MPH student, Hamdard University Bangladesh
Locations (1):
- Hamdard University Bangladesh, Munshiganj, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting 6 months after publication.
Access Criteria: Request by email.